CLINICAL TRIAL: NCT07303088
Title: Effects of L-Carnitine and Coenzyme Q10 Supplementation on Oxidative Stress in Tunisian Hemodialysis Patients: The L-Car-Q10 Study-A Randomized Clinical Trial.
Brief Title: Effects of L-carnitine and Coenzyme Q10 Supplementation on Oxidative Stress in Tunisian Hemodialysis Patients.
Acronym: L-car-Q10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sfax (Other)
Responsible Party: Principal Investigator, Azza KHEDHIRI, MD, Head of hemodialysis unit, Sfax CNSS polyclinic, University of Sfax
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 31/24
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Oxidative Stress Response; Hemodialysis; End Stage Kidney Disease (ESRD)
Keywords: oxidative stress; end stage kidney disease (ESRD); hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Carnitine; coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- L-carnitine group (Active Comparator): L-carnitine group: 18 patients, receiving oral supplementation of 1000Mg of L-carnitine (two capsules of 500 mg of L-carnitine each), and one placebo capsule identical to Coenzyme Q10.
  Interventions: Dietary Supplement: Oral administration of L-carnitine 1000 Mg
- Coenzyme Q10 group (Active Comparator): Coenzyme Q10 group: 19 patients, receiving one capsule of 300 mg of Q10, and two placebo capsules identical to L-carnitine
  Interventions: Dietary Supplement: Oral administration of Coenzyme Q10 300Mg
- Placebo group (Placebo Comparator): Placebo group: 15 patients, receiving two placebo capsules identical to L-carnitine and one placebo capsule identical to Coenzyme Q10
  Interventions: Other: placebo capsules
- Control group (No Intervention): a group of 34 healthy subjects collected from the regional blood transfusion center, with no systemic or chronic disease.

INTERVENTIONS:
Dietary Supplement: Oral administration of L-carnitine 1000 Mg — Oral administration of 1000mg of L-carnitine per day ( two oral capsules of 500mg) in L-carnitine group, and one placebo capsule identical to Coenzyme Q10.
  Other Names: two capsules of 500Mg of L-carnitine
  Arms: L-carnitine group
Dietary Supplement: Oral administration of Coenzyme Q10 300Mg — Oral administration of 300mg of Coenzyme Q10 per day (one oral capsule of 300mg) in Coenzyme Q10 group, with two placebo capsules identical to L-carnitine.
  Other Names: one capsule of 300Mg of Coenzyme Q10
  Arms: Coenzyme Q10 group
Other: placebo capsules — Oral administration of placebos: Two placebo capsules identical to L-carnitine and one placebo capsule identical to Coenzyme Q10 tablets.
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial was to learn if supplementation with L-carnitine or Coenzyme Q10 improves effectively the oxidative stress markers in adult patients undergoing chronic hemodialysis. It was also to evaluate the basic oxidative profile of hemodialyzed patients and to learn about the safety and tolerability of the two supplements. The main questions it aimed to answer are:

* Does tunisian hemodialyzed patients have a severe oxidative status?
* Does L-carnitine and Coenzyme Q10 significantly reduce oxidant markers and improve endogenous antioxidants compared to placebo?
* Are the positive effects of L-carnitine and Coenzyme Q10 on oxidative stress maintained after a period of wash-out ?
* Are L-carnitine and Coenzyme Q10 supplementation safe and well-tolerated in hemodialyzed patients?

Researchers had compared the effects of the two supplements to identical placebos. Oxidative parameters were dosed at baseline, after 12 weeks of supplementation, and after 12 weeks of wash-out. Participants had:

* taken one of the active molecules or a placebo for 12 weeks.
* been followed-up for 12 more weeks of wash-out after the end of the cure.
* a monitoring by hebdomadary sheets in each hemodialysis session, that recorded the medication taken the day of the hemodialysis session and the day before, errors and forgetfulness of the medication, as well as any incidents or adverse events, and monthly visits to monitor patient safety, compliance, and collect key clinical data including blood pressure, dry weight, and specific laboratory tests like hemoglobin and thyroid function, all of which were recorded in the Case Report Form (CRF).

DETAILED DESCRIPTION:
The study design was a prospective, randomized, double-blind, and placebo-controlled clinical trial, aiming to compare the effects of the two active molecules to identical-looking placebos. After a visit of pre-selection, elligible Patients were randomly assigned to one of the three intervention groups (L-car, Q10, or placebo), using a computer-generated list of random numbers. The target population comprised adult patients aged between 18 and 85 years, with end-stage renal disease, undergoing chronic hemodialysis for more than 6 months, with high-flux dialyzers, and receiving an adequate dialysis dose with satisfactory uremia control. Strict exclusion criteria included patients' history of poor medication adherence, severe intercurrent infection, hepatocellular failure, or a recent major cardiovascular event, or those receiving antioxidant treatment within one to six months before the study, depending on the type of antioxydant. The treatment course lasted 12 weeks and consisted of: (i) L-carnitine group: Two capsules of 500 mg of L-car each, and one placebo capsule identical to Q10; (ii) Coenzyme Q10 group: One capsule of 300 mg of Q10, and two placebo capsules identical to L-car; and (iii) Placebo group: Two placebo capsules identical to L-car and one placebo capsule identical to Q10. Plasma levels of malondialdehyde (MDA), advanced oxidation protein products (AOPP), vitamin C, and glutathione (GSH), as well as the activities of superoxide dismutase (SOD), catalase (CAT), and glutathione peroxidase (Gpx), were measured in plasma by spectrophotometry before treatment, after the 12-week course, and following a 12-week washout period.

In addition to the study groups, a group of 34 healthy subjects (control group) was collected. The same parameters were measured in this group to evaluate the baseline oxidative status of HD group. The study protocol received approval from the local ethics committee before the initiation of any recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Patients on chronic hemodialysis for at least 6 months.
* Age between 18 and 85 years old.
* Chronic hemodialysis performed 3 times per week with high-flux dialyzers.
* Adequate dialysis dose : PRU ≥ 65% and/or KT/V > 1.1.
* Satisfactory control of uremia.
* Life expectancy greater than 1 year.

Exclusion Criteria:

* History of Poor medication adherence.
* Severe intercurrent infection.
* Severe hepatocellular insufficiency.
* Major cardiovascular event within 3 months before the study.
* Intake of antioxidants (except vitamin D2 and/or active vitamin D).
* Intake of vitamins E, D3, or B9 → Washout period of at least 1 month.
* Intake of L-car, other amino acids, or CoQ10 → Washout period of at least 6 months.
* Withdrawal of consent.
* Major digestive intolerance/adverse effect during the intervention.
* Severe infection/major cardiovascular event during the study.
* Patient refusal to continue the trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Oxidative stress parameters | T1: Before Treatment; T2: At the end of the 12-week course; T3: After 12 weeks of wash-out
  Plasma levels of malondialdehyde (MDA), advanced oxidation protein products (AOPP), vitamin C, and glutathione (GSH), as well as the activities of superoxide dismutase (SOD), catalase (CAT), and glutathione peroxidase (Gpx), were measured in plasma by spectrophotometry before treatment, after the 12-week course, and following a 12-week washout period.

CONTACTS AND LOCATIONS:
Overall Officials: Lobna Ben Mahmoud, MD, PhD, Medicine professor, Study Director — University of Sfax
Locations (1):
- Social security fund polyclinic, Sfax, Sfax Ville, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Raw results of the various measured parameters in Excel files, the informed consent model, the CRF model, and the follow-up sheets models, once the article is officially accepted for publication. The datasets analyzed during the study are available from the corresponding author on reasonable request
Supporting Information: Study Protocol, ICF, CSR
Time Frame: From the date of publication of the article and for a limited duration of 5 years.
Access Criteria: Qualified researchers and authorized personnel who have received formal approval for a secondary use proposal. They would be able to access relevant study documentation such as the study protocol, the Statistical Analysis Plan (SAP), the informed consent model and the blank Case Report Forms (CRFs).Approved researchers must sign a formal Data Sharing Agreement (DSA) that outlines strict conditions for data usage, prohibiting any attempt to re-identify participants.